CLINICAL TRIAL: NCT05710835
Title: Application Study of Infusing Irritant Medications Through Midline Catheter Based on Real World Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sir Run Run Shaw Hospital (Other)
Responsible Party: Principal Investigator, Zhao Linfang, assitant nursing director, Sir Run Run Shaw Hospital
Other Study IDs: IVTEAM202301
Record Dates: First submitted 2023-01-04; First posted 2023-02-02 (Actual); Last update posted 2023-02-02 (Actual); Status verified 2023-01

CONDITIONS: Catheter Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- irritant medications group: Patients who used midline catheter to infuse irritant medications.
- nonirritant medications group: Patients who used midline catheter to infuse nonirritant medications.

SUMMARY:
The goal of this observational study is to learn about the effect on midline catheter outcomes when infusing irritant medications through midline catheter. The main questions it aims to answer are:Identify the current situation of infusing irritant medications through midline catheter;Explore the effect on midline catheter outcomes when infusing irritant medications through midline catheter;Identify specific medications that affect catheter outcomes.

DETAILED DESCRIPTION:
First, the patients were divided into two groups according to whether irritant medications were infused or not,then observed the rate of complications between the two groups.Second, grouped according to the irritant medications, Identify specific medications that affect catheter outcomes through statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥14 years old
* Patients who had a midline catheter

Exclusion Criteria:

* Patients who received vesicant medications through the midline catheter
* Patients who had both a midline catheter and a central vascular access device

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients at a 3A hospital
Sampling Method: Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
catheter complications | during catheter indwelling
  catheter complications rate

CONTACTS AND LOCATIONS:
Overall Officials: Linfang Zhao, Principal Investigator — Sir Run Run Shaw Hospital
Locations (1):
- Linfang Zhao, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Adams DZ, Little A, Vinsant C, Khandelwal S. The Midline Catheter: A Clinical Review. J Emerg Med. 2016 Sep;51(3):252-8. doi: 10.1016/j.jemermed.2016.05.029. Epub 2016 Jul 5. PMID 27397766
- [Background] Qin KR, Pittiruti M, Nataraja RM, Pacilli M. Long peripheral catheters and midline catheters: Insights from a survey of vascular access specialists. J Vasc Access. 2021 Nov;22(6):905-910. doi: 10.1177/1129729820966226. Epub 2020 Oct 20. PMID 33078685
- [Background] Gorski LA, Hadaway L, Hagle ME, Broadhurst D, Clare S, Kleidon T, Meyer BM, Nickel B, Rowley S, Sharpe E, Alexander M. Infusion Therapy Standards of Practice, 8th Edition. J Infus Nurs. 2021 Jan-Feb 01;44(1S Suppl 1):S1-S224. doi: 10.1097/NAN.0000000000000396. No abstract available. PMID 33394637
- [Background] Prasanna N, Yamane D, Haridasa N, Davison D, Sparks A, Hawkins K. Safety and efficacy of vasopressor administration through midline catheters. J Crit Care. 2021 Feb;61:1-4. doi: 10.1016/j.jcrc.2020.09.024. Epub 2020 Oct 2. PMID 33049486
- [Background] Anderson J,Greenwell A,Louderback J,et al.Comparison of Outcomes of Extended Dwell/Midline Peripheral Intravenous Catheters and Peripherally Inserted Central Catheters in Children[J].Journal of Vascular Access,2016,21(3): 158-164.
- [Background] Knottnerus JA, Tugwell P. Real world research. J Clin Epidemiol. 2010 Oct;63(10):1051-2. doi: 10.1016/j.jclinepi.2010.08.001. No abstract available. PMID 20728043
- [Background] Mermel LA, Parenteau S, Tow SM. The risk of midline catheterization in hospitalized patients. A prospective study. Ann Intern Med. 1995 Dec 1;123(11):841-4. doi: 10.7326/0003-4819-123-11-199512010-00005. PMID 7486466
- [Background] Hallam C, Weston V, Denton A, Hill S, Bodenham A, Dunn H, Jackson T. Development of the UK Vessel Health and Preservation (VHP) framework: a multi-organisational collaborative. J Infect Prev. 2016 Mar;17(2):65-72. doi: 10.1177/1757177415624752. Epub 2016 Jan 10. PMID 28989456
- [Background] Alexandrou E,Ramjan LM,Spencer T,et al.The use of midline catheters in the adult acute care setting-clinical implications and recommendations for practice[J]. Journal of the Association for Vascular Access,2011,16(1): 35-41.
- [Background] Marsh N, Webster J, Larson E, Cooke M, Mihala G, Rickard CM. Observational Study of Peripheral Intravenous Catheter Outcomes in Adult Hospitalized Patients: A Multivariable Analysis of Peripheral Intravenous Catheter Failure. J Hosp Med. 2018 Feb 1;13(2):83-89. doi: 10.12788/jhm.2867. Epub 2017 Oct 18. PMID 29073316
- [Background] Anderson NR. Midline catheters: the middle ground of intravenous therapy administration. J Infus Nurs. 2004 Sep-Oct;27(5):313-21. doi: 10.1097/00129804-200409000-00005. PMID 15385895
- [Background] O'Grady NP, Alexander M, Burns LA, Dellinger EP, Garland J, Heard SO, Lipsett PA, Masur H, Mermel LA, Pearson ML, Raad II, Randolph AG, Rupp ME, Saint S; Healthcare Infection Control Practices Advisory Committee. Guidelines for the prevention of intravascular catheter-related infections. Am J Infect Control. 2011 May;39(4 Suppl 1):S1-34. doi: 10.1016/j.ajic.2011.01.003. No abstract available. PMID 21511081
- [Background] Mushtaq A, Navalkele B, Kaur M, Krishna A, Saleem A, Rana N, Gera S, Chandramohan S, Surapaneni M, Chopra T. Comparison of complications in midlines versus central venous catheters: Are midlines safer than central venous lines? Am J Infect Control. 2018 Jul;46(7):788-792. doi: 10.1016/j.ajic.2018.01.006. Epub 2018 Mar 7. PMID 29525366
- [Background] DeVries M, Lee J, Hoffman L. Infection free midline catheter implementation at a community hospital (2 years). Am J Infect Control. 2019 Sep;47(9):1118-1121. doi: 10.1016/j.ajic.2019.03.001. Epub 2019 Apr 30. PMID 31047692
- [Background] Sharp R, Esterman A, McCutcheon H, Hearse N, Cummings M. The safety and efficacy of midlines compared to peripherally inserted central catheters for adult cystic fibrosis patients: a retrospective, observational study. Int J Nurs Stud. 2014 May;51(5):694-702. doi: 10.1016/j.ijnurstu.2013.09.002. Epub 2013 Sep 14. PMID 24103730
- [Background] Lisova K, Hromadkova J, Pavelkova K, Zauska V, Havlin J, Charvat J. The incidence of symptomatic upper limb venous thrombosis associated with midline catheter: Prospective observation. J Vasc Access. 2018 Sep;19(5):492-495. doi: 10.1177/1129729818761276. Epub 2018 Mar 16. PMID 29546782
- [Background] Dickson HG, Flynn O, West D, Alexandrou E, Mifflin N, Malone M. A Cluster of Failures of Midline Catheters in a Hospital in the Home Program: A Retrospective Analysis. J Infus Nurs. 2019 Jul/Aug;42(4):203-208. doi: 10.1097/NAN.0000000000000330. PMID 31283663
- [Background] Cawcutt KA, Hankins RJ, Micheels TA, Rupp ME. Optimizing vascular-access device decision-making in the era of midline catheters. Infect Control Hosp Epidemiol. 2019 Jun;40(6):674-680. doi: 10.1017/ice.2019.49. Epub 2019 Mar 29. PMID 30924436
- [Background] Nielsen EB, Antonsen L, Mensel C, Milandt N, Dalgaard LS, Illum BS, Arildsen H, Juhl-Olsen P. The efficacy of midline catheters-a prospective, randomized, active-controlled study. Int J Infect Dis. 2021 Jan;102:220-225. doi: 10.1016/j.ijid.2020.10.053. Epub 2020 Oct 28. PMID 33129962
- [Background] Elli S, Pittiruti M, Pigozzo V, Cannizzo L, Giannini L, Siligato A, Rondelli E, Foti G, Lucchini A. Ultrasound-guided tip location of midline catheters. J Vasc Access. 2020 Sep;21(5):764-768. doi: 10.1177/1129729820907250. Epub 2020 Feb 28. PMID 32106761
- [Background] Caparas JV, Hu JP. Safe administration of vancomycin through a novel midline catheter: a randomized, prospective clinical trial. J Vasc Access. 2014 Jul-Aug;15(4):251-6. doi: 10.5301/jva.5000220. Epub 2014 Apr 8. PMID 24811603